CLINICAL TRIAL: NCT05494658
Title: A Multicenter Randomized Controlled Study of Preoperative Oral Administration of Branched-chain Amino Acids in Reducing Postoperative Insulin Resistance in Colorectal Cancer Patients
Brief Title: Impact of Preoperative Oral Branched-chain Amino Acids on Reducing Postoperative Insulin Resistance.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Peng (Other)
Collaborators: Huashan Hospital (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor-Investigator, Sun Peng, Executive Director of General Surgery, Shanghai Tong Ren Hospital
Organization: Shanghai Tong Ren Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-050-01
Record Dates: First submitted 2022-07-26; First posted 2022-08-10 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Insulin Resistance; Colorectal Cancer
Keywords: postoperative insulin resistance; branched chain amino acids; colorectal cancer
MeSH Terms: conditions — Insulin Resistance; Colorectal Neoplasms | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- research group (Experimental): 600ml drink which contains 18g BCAA was consumed by patients 2-4h before surgery.
  Interventions: Dietary Supplement: BCAA
- control group (Placebo Comparator): 600ml water was consumed by patients 2-4h before suegery.
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: BCAA — 600ml drink which contains 18g BCAA was consumed by patients 2-4h before surgery.
  Arms: research group
Dietary Supplement: water — 600ml water was consumed by patients 2-4h before suegery.
  Arms: control group

SUMMARY:
Postoperative insulin resistance refers to the phenomenon that the body's glucose uptake stimulated by insulin is reduced due to stress effects such as trauma or the inhibitory effect of insulin on liver glucose output is weakened after surgery.

There is a clear link between postoperative insulin resistance and poor perioperative prognosis. Therefore, exploring interventions to reduce postoperative stress insulin resistance, stabilize postoperative blood glucose, and reduce postoperative complications are clinical problems that need to be solved urgently. In recent years, research on branched-chain amino acids and metabolic diseases has become a hot spot. Studies have found that in the rat model, preoperatively given a high branched-chain amino acid diet can inhibit postoperative insulin resistance and stabilize blood glucose levels. This research plan is to try to add branched-chain amino acids before surgery to observe the occurrence of postoperative insulin resistance in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years old ;
2. Clinical diagnosis of colorectal cancer;
3. Planned elective laparoscopic radical resection of colorectal cancer;
4. Preoperative American Society of Anesthesiologists（ASA）score grade I-III ;
5. Informed consent was obtained from patients.

Exclusion Criteria:

1. Clinical diagnosis of Diabetes mellitus;
2. Preoperative insulin resistance ;
3. Renal insufficiency requires dialysis, hepatic insufficiency (Child - Pugh grade B and above);
4. Eating disorders caused by gastrointestinal obstruction;
5. Pregnant or lactating women;
6. Patients with severe mental illness.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of postoperative blood glucose>8mmol/L | 1 day
  The proportion of postoperative blood glucose>8mmol/L.Measure method：Continuous blood glucose meter.

SECONDARY OUTCOMES:
Postoperative blood glucose | 1 day
  Measured by continuous blood glucose meter
Homeostasis model assessment - insulin resistance （HOMA-IR） | 1 day
  Measured by blood test. HOMA-IR = (blood glucose [mmol/L] × blood insulin [μunits/mL])/22.5.
Postoperative complications | 1 month
  Postoperative complications include branched-chain amino acid-related complications, surgery-related complications, and systemic complications. Postoperative complications were graded according to the Clavien-Dindo system
Postoperative hospital stay | 1 month
  Postoperative hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongren Hospital, Shanghai, China